CLINICAL TRIAL: NCT07231367
Title: "Cholesterol-lowering Potential of Sunflower Seeds: Evidence From Phytochemical and Fatty Acid Composition and a Randomized Human Trial"
Brief Title: Effect of Sunflower Seed Consumption on Blood Cholesterol Levels in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Faisalabad (Other)
Responsible Party: Principal Investigator, Amna Butt, Lecturer, University of Faisalabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUNSEED-CHOL
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Hypercholesterolemia
Keywords: Sunflower seeds; Hypercholesterolemia; Cholesterol; Phytochemicals
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants continued their usual diet without consuming sunflower seeds. Blood cholesterol and lipid profiles were measured at baseline and at the end of the study period.
- Diseased Group (Experimental): Participants consumed a defined daily portion of sunflower seeds for the duration of the study. Blood samples were collected at baseline and after the intervention to measure total cholesterol, LDL-C, HDL-C, triglycerides, and other lipid parameters. Dietary intake and adherence to the intervention were monitored throughout the study period
  Interventions: Dietary Supplement: Sunflower Seed Supplementation

INTERVENTIONS:
Dietary Supplement: Sunflower Seed Supplementation — Participants consumed sunflower seeds daily for 45 days
  Arms: Diseased Group

SUMMARY:
This study evaluates the effect of daily consumption of sunflower seeds on blood cholesterol levels in adult participants. Participants were randomly assigned to consume a specified amount of sunflower seeds for a defined period, and their blood cholesterol and lipid profile were measured before and after the intervention. The study aims to determine whether sunflower seeds can contribute to improving cardiovascular health by lowering cholesterol. Adult men and women meeting the eligibility criteria were included in the study. The findings may help inform dietary recommendations for managing cholesterol and promoting heart health.

DETAILED DESCRIPTION:
This randomized, open-label human trial evaluated the cholesterol-lowering potential of sunflower seeds in adult participants. Eligible men and women were recruited based on inclusion criteria, which included age range, baseline cholesterol levels, and absence of major health conditions. Participants were randomly assigned to consume a defined daily portion of sunflower seeds for a specified intervention period. Blood samples were collected at baseline and at the end of the intervention to measure total cholesterol, LDL-C, HDL-C, triglycerides, and other relevant lipid parameters.

Prior to the human intervention, sunflower seeds were analyzed for their nutritional composition, mineral content, phytochemical profile, and fatty acid composition using standard laboratory procedures. Tests included proximate analysis (moisture, protein, fat, ash, and carbohydrate content), mineral quantification (calcium, magnesium, potassium, etc.), phytochemical assays (total phenolics, flavonoids), and fatty acid profiling using gas chromatography. These analyses provided a detailed characterization of the seeds' bioactive components relevant to cardiovascular health.

The study also included assessments of dietary intake, anthropometric measurements, and adherence to the intervention. The primary objective was to determine the effect of sunflower seed consumption on blood cholesterol levels, while secondary objectives included evaluating changes in lipid profile and potential associations with bioactive components of the seeds. Data were analyzed using standard statistical methods. The results aim to provide evidence on the role of sunflower seeds in cardiovascular risk management and to inform dietary recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Participants included males aged between 40 and 50 years, with serum cholesterol levels exceeding 200 mg/dL, and shared the same socioeconomic status.

Exclusion Criteria:

* The participants were excluded based on different physiological factors, such as active smokers, alcoholics, chronic disease patients, people having extremely low or high BMI, people suffering from psychological disorders or familial hypercholesterolemia, people who belong to a high-income group, and people having doubts or confusion while following instructions

Ages: 40 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2023-08-20 (Actual); Study Completion 2023-08-20 (Actual)

PRIMARY OUTCOMES:
Change in Total Cholesterol | Baseline and 45 days after intervention
  Total serum cholesterol measured using standard enzymatic methods at baseline and at the end of the 45 days sunflower seed supplementation period.

SECONDARY OUTCOMES:
LDL Cholesterol | Baseline and 45 days after intervention
  LDL cholesterol measured using standard enzymatic methods at baseline and at the end of the 45 days supplementation period.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Agriculture, Faisalabad, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
The study was completed prior to an IPD sharing plan, and participant consent did not include sharing of individual-level data.